CLINICAL TRIAL: NCT03393299
Title: Impact of the Systematic Use of the Criteria STOPP/START in Short Stay Geriatric: Study of Superiority, Randomized, Controlled, Prospective, Single Blind
Brief Title: Impact of the Systematic Use of the Criteria STOPP/START in Short Stay Geriatric.
Acronym: REVOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RC-P0059
Record Dates: First submitted 2018-01-02; First posted 2018-01-08 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Quality of Life; Drug Use
Keywords: elderly people; geriatric short-stay; STOPP/START criteria
MeSH Terms: interventions — Potentially Inappropriate Medication List

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STOPP/START (Experimental): Use of STOPP/START criteria during medication reconciliation
  Interventions: Procedure: STOPP/START criteria
- CONTROL (No Intervention): Medication reconciliation done as usual, without the consideration of the STOPP/START criteria

INTERVENTIONS:
Procedure: STOPP/START criteria — software which helps to do the drug reconciliation
  Arms: STOPP/START

SUMMARY:
Assess the impact of the systematic use of STOPP/START tool during medication conciliation on the evolution of hospitalised elderly people's quality of life at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with more than 75 years old
* Hospitalized in geriatrics short-stay
* Patient with a written informed consent
* Patient with a social security scheme

Exclusion Criteria:

* Severe dementia
* Not able to respond to SF-12
* Disease at final stage
* Patient under legal protection (maintenance of justice, tutelage, legal guardianship)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
SF-12 Quality of life scale | at inclusion and at 2 months
  The evolution of the hospitalised elderly people's quality of life at 2 months will be measured by the SF-12 scale.

SECONDARY OUTCOMES:
Number of falls | at 2 months
  The number of falls during the two months following the inclusion will be collected for each patient.
Proportion of patients rehospitalized | at 2 months
  The proportion of patients that have been rehospitalized (unscheduled hospitalization) during the two months following inclusion will be measured.
Mortality | at 2 months
  The mortality during the two months following inclusion will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital La Porte Verte, Versailles, France

IPD SHARING:
Plan to Share IPD: No